CLINICAL TRIAL: NCT05028764
Title: A Study to Determine the Range of Tissue Frataxin Concentrations and Other Potential Biomarkers for Friedreich's Ataxia in Normal Healthy Volunteers
Brief Title: Determine Range of Tissue Frataxin Concentrations and Other Potential Biomarkers
Status: Completed | Type: Observational
Sponsor: Larimar Therapeutics, Inc. (Industry)
Collaborators: Clinilabs, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: CLIN-1601-002
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Friedreich Ataxia; Healthy Volunteers
MeSH Terms: conditions — Friedreich Ataxia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal cells and blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 18 to 30 years of age group: Consisting of at least 13 males and 13 females
  Interventions: Diagnostic Test: Buccal Swabs, Blood Draws and Skin Punch Biopsy
- 31 to 50 years of age group: Consisting of at least 13 males and 13 females
  Interventions: Diagnostic Test: Buccal Swabs, Blood Draws and Skin Punch Biopsy

INTERVENTIONS:
Diagnostic Test: Buccal Swabs, Blood Draws and Skin Punch Biopsy — Buccal Swabs - FXN and specific RNA markers; Blood Draws - Lipid panel, Protein Marker Analysis and Gene RNA Analysis; Skin Punch Biopsy - Protein Markers

SUMMARY:
To examine range of tissue frataxin (FXN) concentrations, specific ribonucleic acids, other proteins and specialized lipids in the buccal cells, blood, and skin cells of normal healthy volunteers without Friedreich's ataxia (FRDA).

DETAILED DESCRIPTION:
Primary Objective: To examine the range of tissue frataxin (FXN) concentrations in the buccal cells, blood, and skin cells of normal healthy volunteers without FRDA.

Secondary Objective: To examine the range of specific ribonucleic acids (RNAs), other proteins, and specialized lipids in the buccal cells, blood, and skin cells of normal healthy volunteers without FRDA.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy male or female,18-50 years of age
2. Subject has a body mass index (BMI) ≥18.0 and ≤32.0 as of the screening visit.
3. Subject is racially Caucasian, Asian, Native Hawaiian, or Native American.

Exclusion Criteria:

1. Subject used erythropoietin, etravirine, or gamma interferon within 3 months prior to the Day 1 (assessment) visit.
2. Subject has a chronic condition that requires ongoing prescription drug treatment.
3. Subject use of any statin medications within 3 months before the Day 1 (assessment) visit.
4. Subject use of any lipid-lowering agents, other than statins, within 6 weeks before the Day 1 (assessments) visit.
5. Subject is racially black or African American.
6. Pregnant or breast-feeding female subjects.
7. Subject has a known history of drug or alcohol abuse or current suspected drug or alcohol abuse.
8. Subject is positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg), or hepatitis A virus (HAV).
9. Subject has any condition, disease, or situation, that in the opinion of the principal investigator (PI), could confound the results of the study or put the subject at undue risk, making participation inadvisable.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Examine tissue frataxin concentrations in buccal cells, blood and skin cells | 1 day
  Range of tissue frataxin levels in buccal cells, blood and skin cells

SECONDARY OUTCOMES:
Examine specific ribonucleic acids (RNAs), other proteins, and specialized lipids in buccal cells and blood | 1 day
  Range of specific ribonucleic acids (RNAs), other proteins, and specialized lipids in buccal cells and blood

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Shenouda, M.D., Principal Investigator — Clinilabs, Inc.
Locations (1):
- Clinilabs Drug Development Corporation, Eatontown, New Jersey, United States

REFERENCES:
- [Background] Deutsch EC, Santani AB, Perlman SL, Farmer JM, Stolle CA, Marusich MF, Lynch DR. A rapid, noninvasive immunoassay for frataxin: utility in assessment of Friedreich ataxia. Mol Genet Metab. 2010 Oct-Nov;101(2-3):238-45. doi: 10.1016/j.ymgme.2010.07.001. Epub 2010 Jul 8. PMID 20675166